CLINICAL TRIAL: NCT04221906
Title: A Phase Ib, Multi-Center, Randomized, Vehicle- and Comparator-Controlled Trial, Double-Blind for the Investigational Medicinal Products, Observer-Blind for the Comparators to Evaluate the Safety and Antipsoriatic Efficacy of BOS-475 in a Psoriasis Plaque Test
Brief Title: Study to Evaluate the Safety and Antipsoriatic Efficacy of BOS-475 in a Psoriasis Plaque Test
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BOS-475-102; 2019-002447-17 (EudraCT Number)
Record Dates: First submitted 2020-01-07; First posted 2020-01-09 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Chronic Plaque Psoriasis
Keywords: BOS-475; antipsoriatic efficacy; safety; psoriasis plaque test

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- BOS-475 0.5% (Experimental): Daily application of BOS-475 0.5%
  Interventions: Drug: BOS-475
- BOS-475 1% (Experimental): Daily application of BOS-475 1%
  Interventions: Drug: BOS-475
- BOS-475 2% (Experimental): Daily application of BOS-475 2%
  Interventions: Drug: BOS-475
- Active ingredient-free vehicle cream (Placebo Comparator): Daily application of vehicle cream
  Interventions: Drug: Active ingredient-free vehicle cream
- Daivonex cream (Active Comparator): Daily application of Daivonex cream (calcipotriol 0.005%)
  Interventions: Drug: Daivonex cream (calcipotriol 0.005%)
- Betnesol-V cream (betamethasone 0.1%) (Active Comparator): Daily application of Betnesol-V cream (betamethasone 0.1%)
  Interventions: Drug: Betnesol-V cream (betamethasone 0.1%)

INTERVENTIONS:
Drug: BOS-475 — topical cream
  Arms: BOS-475 0.5%; BOS-475 1%; BOS-475 2%
Drug: Active ingredient-free vehicle cream — topical cream
  Arms: Active ingredient-free vehicle cream
Drug: Daivonex cream (calcipotriol 0.005%) — topical cream
  Arms: Daivonex cream
Drug: Betnesol-V cream (betamethasone 0.1%) — topical cream
  Arms: Betnesol-V cream (betamethasone 0.1%)

SUMMARY:
This study is being conducted to evaluate the safety of topical BOS-475 compared to topically applied comparator formulations and vehicle.

DETAILED DESCRIPTION:
This is a three-center, randomized, placebo- and comparator-controlled, double-blind for the Investigational Medicinal Products (IMPs), observer-blind for the controls, intraindividual comparison of all 6 treatments.

ELIGIBILITY:
Inclusion Criteria:

* Men, or women of non-childbearing potential aged 18-69 years (inclusive)
* Participants with chronic stable plaque psoriasis
* The target lesion(s) should be on the trunk or extremities (excluding palms/soles); psoriatic lesions on the knees or elbows are not to be used as target lesions.
* Willing and able to follow all trial procedures and complete the whole trial
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the Informed Consent Form (ICF) and in this protocol
* Willing to refrain from using any topical treatments on the target areas, other than those mandated by the protocol or for protocol procedures

Exclusion Criteria:

* Other skin disease or infection that is considered by the investigator to be relevant to the outcome of the trial
* Participants with acute psoriasis guttata, psoriasis punctata, psoriasis erythrodermatica or pustular psoriasis
* Any topical antipsoriatics on plaques potentially to be treated in this trial (including corticosteroids, vitamin D analogues, immunomodulators, retinoids, dithranol and tar) in the 4 weeks before first treatment and/or during the trial (pretreatment with salicylic acid is permitted on selected plaques; treatment on the face, ears and scalp is also permitted as lesions are not involved in the trial)
* Systemic treatment with antipsoriatics, e.g., corticosteroids, cytostatics, retinoids, dimethylfumarate or apremilast in the three months before first treatment and during the trial
* Systemic treatment with biological treatments: ustekinumab or secukinumab within six months or adalimumab, infliximab, and etanercept within three months before first treatment and during the trial. Any other previously used biologics for treatment of psoriasis should have been washed out for five half lives before first treatment.
* Ultraviolet A (UVA) or B-therapy within four weeks and psoralen and ultraviolet A (PUVA)-therapy within eight weeks before first treatment and during the trial treatment with concomitant medication that may affect and provoke or aggravate psoriasis, e.g., antimalarial drugs, lithium, beta-blockers, or angiotensin-converting-enzyme (ACE) inhibitors unless on a stable dose for 3 months before trial medication initiation
* History of malignancy within 5 years prior to dosing, except adequately treated non-invasive skin cancer (basal or squamous cell carcinoma
* Positive urine drug or breath alcohol test results during screening or at Day 1, or history of drug abuse within a year prior to the screening visit
* Excess alcohol consumption within 6 months prior to the trial defined as an average weekly intake of > 14 units for males and females. One unit is equivalent to 8 grams of alcohol: a half-pint (~240 milliliters [mL]) of beer, 1 glass (125 mL) of wine, or 1 (25 mL) measure of spirits
* Blood pressure (BP) >160 millimeters of mercury (mmHg) systolic or >95 mmHg diastolic at screening
* Participation in another clinical trial within the last six months for biological agents, or four weeks for small molecules prior to first treatment in this clinical trial

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
Number of treatment-emergent adverse events (TEAEs) | up to Day 19
Number of treatment-emergent application site reactions | up to Day 19
Change from Baseline in systolic and diastolic blood pressure | Baseline; up to Day 19
Change from Baseline in pulse | Baseline; up to Day 19
Change from Baseline in respiration | Baseline; up to Day 19
Change from Baseline in body temperature | Baseline; up to Day 19
Number of participants with clinically significant physical examination findings | up to Day 19

SECONDARY OUTCOMES:
Change from Baseline in psoriatic infiltrate thickness on Day 19 (assessed by measurement of the thickness of the Echo Poor Band [EPB] of the inflammatory infiltrate using 22-megahertz (MHz) sonography) | Baseline; Day 19
Change from Baseline in psoriatic infiltrate thickness on Days 8 and 15 (assessed by measurement of the thickness of the EPB of the inflammatory infiltrate using 22-MHz sonography) | Baseline; Days 8 and 15
Area under the curve (AUC) of change from Baseline in thickness of the EPB of the inflammatory infiltrate | Baseline; Day 19
Change from Baseline in the test fields compared to the surrounding plaque skin, as an evaluation of the antipsoriatic efficacy by clinical assessment, using a 5-point score | Baseline; Days 1, 8, 15, and 19 (End of Trial)
  -1 = worsened; 0 = unchanged (no effect); 1 = slight improvement; 2 = clear improvement but not completely healed; 3 = completely healed.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaobing Qian, MD, PhD, Study Director — Boston Pharmaceuticals, Vice President, Clinical Development
Locations (3):
- Germany (3):
  - Gemeinschaftspraxis Dr. med. Johannes Niesmann und Dr. med. Nick Othlinghaus Hauszentrum im Jahrhunderthaus - Zentrum für klinische Studien, Bochum
  - bioskin GmbH, Hamburg
  - Klinische Forschung Schwerin GmbH, Schwerin

IPD SHARING:
Plan to Share IPD: No